CLINICAL TRIAL: NCT06324461
Title: Glucagon-like Peptide-1 Receptor Agonist for Reduction of Myocardial Injury After Non-Cardiac Surgery
Brief Title: GLP-1 Receptor Agonist for Reduction of Myocardial Injury After Non-cardiac Surgery
Acronym: GLUMINS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Research Grants Council, Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Chun Ka, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GLUMINS
Record Dates: First submitted 2023-03-30; First posted 2024-03-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Myocardial Injury
Keywords: Myocardial injury following non-cardiac surgery; glucagon-like peptide 1 receptor agonists; Dulaglutide
MeSH Terms: interventions — dulaglutide; Injections, Subcutaneous

STUDY DESIGN:
Intervention Model Description: Open-labelled, superiority randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dulaglutide group (Experimental): Subject randomized into this group will receive single subcutaneous dose of Dulaglutide 0.75mg 1 to 14 days prior to surgery, on top of routine peri-operative care
  Interventions: Drug: Dulaglutide 0.75mg subcutaneous injection
- Control group (No Intervention): Subject randomized into this group will receive routine peri-operative care

INTERVENTIONS:
Drug: Dulaglutide 0.75mg subcutaneous injection — Subject randomized into treatment group will receive single subcutaneous dose of Dulaglutide 0.75mg 1 to 14 days prior to surgery
  Other Names: Trulicity 0.75mg subcutaneous injection
  Arms: Dulaglutide group

SUMMARY:
This is an investigator initiated, multi-center, open-labelled, superiority randomized controlled trial of 372 patients undergoing elective non-cardiac surgery. Recruited patients will be randomized in a 2:1 ratio to receive single subcutaneous dose of Glucagon-like Peptide-1 Receptor Agonist (GLP-1 RAs) 1 to 14 days prior to surgery or receive routine care.

Dulaglutide (Trulicity; Eli Lilly, USA) is chosen as GLP-1 Receptor Agonists investigational drug for this study. Apart from peri-operative routine care, all recruited subjects will undergo physical, respiratory and cardiac assessments including electrocardiography and blood check including cardiac enzymes. Myocardial injury, cardiovascular outcomes and safety will be assessed and evaluated for efficacy and safety of this prophylactic measurement for the reduction of myocardial injury after non-cardiac surgery.

DETAILED DESCRIPTION:
Myocardial injury following non-cardiac surgery (MINS) is increasingly recognized as a major cause of peri-operative morbidity and mortality worldwide. MINS is defined as post-operative cardiomyocyte injury that can be detected by high-sensitive troponin assays, which may or may not be associated with symptoms or changes on electrocardiogram (ECG). Globally, it was found that 35.5% patients had MINS with elevated troponin level in the early post-operative period. Post-operative troponin T level strongly correlated with peri-operative mortality. It was demonstrated that elevated troponin T level to 14-20 ng/L after surgery significantly increased 30-day mortality with hazard ratio of 9.11. As the global volume of non-cardiac surgeries continues to increase, there is an urgent need to identify effective strategies to minimize MINS. To date, no pharmacological intervention has been shown to safely reduce MINS.

This study will evaluate the effect of pre-operative glucagon-like peptide 1 receptor agonists (GLP-1 RAs) on MINS. GLP-1 is a peptide hormone produced by intestinal epithelial endocrine L-cells that stimulates insulin secretion and inhibits glucagon secretion. GLP-1 RAs have been used to treat both diabetic and non-diabetic conditions. In landmark cardiovascular outcome trials, GLP-1 RAs were shown to reduce major adverse cardiovascular events (MACE) when compared with placebo. GLP-A RAs exert beneficial effects by stabilizing atherosclerotic plaques. Animal studies revealed that a GLP-1 RAs attenuate activation and recruitment of monocytes and macrophages to the arterial wall by suppressing expression of interleukin 6 (IL-6), chemokine (C-C motif) ligand 2 (CCL2), vascular cell adhesion molecule 1 (VCAM-1), and E- selectin (SELE). GLP-1 RAs also suppress vascular smooth muscle cell proliferation and migration via the Cyclic adenosine monophosphate (cAMP) or protein kinase A (PKA) pathway. Another key advantage of using GLP-1 RA in the context of surgery is intra-operative stabilization of glycemic level. It is well established that intra-operative hyperglycemia is associated with increased risk of MINS. Prospective studies have revealed that GLP-1 RA infusion during the peri-operative period resulted in better glycemic control among diabetic and non-diabetic patients without significantly increasing hypoglycemia risk.

The "Glucagon-like Peptide-1 Receptor Agonist for Reduction of Myocardial Injury after Non-Cardiac Surgery" (GLUMINS) trial is an investigator initiated, multi-center, open-labelled Randomized Controlled Trial that will determine the effect of pre-operative GLP-1 RAs on MINS. The study hypothesis is that pre-operative GLP-1 RAs will reduce myocardial injury in patients undergoing non-cardiac surgery. Critically needed new knowledge will be generated about the effectiveness of GLP-1 RAs as a peri-operative intervention to reduce MINS, which may fundamentally alter peri-operative management in non-cardiac surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Planned elective intermediate to high risk non-cardiac surgery under general anesthesia
* Anticipated to remain hospitalized for at least one night after surgery
* Voluntarily agrees to participate by providing written informed consent

Exclusion Criteria:

* History of symptomatic hypoglycemia within 1 month of recruitment
* History of pancreatitis
* Diabetic retinopathy
* Personal or family history of medullary thyroid carcinoma (MTC)
* Multiple Endocrine Neoplasia syndrome type 2 (MEN 2)
* Acute coronary syndrome, decompensated heart failure, cardiogenic shock, or myocarditis within 1 month of recruitment
* Stroke or transient ischemic attack within 1 month of recruitment
* Known severe liver disease (Child-Pugh B or C)
* Stage 5 chronic kidney disease (estimated glomerular filtration rate (eGFR) by Modified Diet in Renal Disease (MDRD) equation < 15 mL/min)
* Recent use of GLP-1 RA within 1 month of recruitment
* Known allergy or hypersensitivity to GLP-1 RA
* Women of childbearing age who are not taking effective contraception, or who are pregnant or breast-feeding
* Use of Dipeptidyl peptidase-4 inhibitor(DPP4i)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with MINS | Within 72 hours after surgery
  Defined as any elevation in troponin T >= 14ng/L

SECONDARY OUTCOMES:
Proportion of patients with composite of non-fatal MINS, non-fatal stroke or cardiovascular mortality | Within 30 days of randomization
Proportion of patients with MINS who do not fulfill the 4th universal definition of myocardial infarction | Within 30 days of randomization
Proportion of patients with myocardial infarction according to the 4th universal definition of myocardial infarction | Within 30 days of randomization
Proportion of patients with ischemic stroke | Within 30 days of randomization
Proportion of patients with cardiovascular death | Within 30 days of randomization
Proportion of patients with all-cause mortality | Within 30 days of randomization
Mean days alive and out of hospital | Within 30 days of randomization
Clinically important atrial fibrillation | Within 30 days of randomization
Clinically significant hypoglycaemia | Within 30 days of randomization
Mean peak troponin T concentration | During the period of index hospitalization up to 3 days
Mean area under curve of troponin T concentration | During the period of index hospitalization up to 3 days

OTHER OUTCOMES:
Proportion of patients with coronary revascularization | Within 30 days of randomization
Proportion of patients who require readmission for cardiovascular conditions | Within 30 days of randomization
Proportion of patients with non-fatal cardiac arrest | Within 30 days of randomization
Proportion of patients who require hospitalization for heart failure | Within 30 days of randomization
Proportion of patients who develop pulmonary embolism and/or deep vein thrombosis | Within 30 days of randomization
Proportion of patients with International Society on Thrombosis and Haemostasis (ISTH) major bleeding | Within 30 days of randomization
Proportion of patients with bleeding independently associated with mortality following noncardiac surgery (BIMS) | Within 30 days of randomization
Proportion of patients with infection or sepsis | Within 30 days of randomization
Proportion of patients with acute renal failure fulfilling Kidney Disease Improving Global Outcomes (KDIGO) criteria | Within 30 days of randomization
Proportion of patients with acute renal failure requiring dialysis | Within 30 days of randomization
Proportion of patients requiring amputation | Within 30 days of randomization
Mean length of stay | During index hospitalization up to 3 days
Mean length of intensive care unit stay | During index hospitalization up to 1 week
Mean days alive without need for intensive care support | During index hospitalization up to 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Chun Ka Wong, Clinical Assistant Professor, Principal Investigator — The University of Hong Kong
Locations (3):
- China (3):
  - Duchess of Kent Children's Hospital at Sandy Bay, Hong Kong, Hong Kong SAR
  - Queen Mary Hospital, Hong Kong, Hong Kong SAR
  - Tung Wah Hospital, Hong Kong, Hong Kong SAR

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Writing Committee for the VSI, Devereaux PJ, Biccard BM, Sigamani A, Xavier D, Chan MTV, Srinathan SK, Walsh M, Abraham V, Pearse R, Wang CY, Sessler DI, Kurz A, Szczeklik W, Berwanger O, Villar JC, Malaga G, Garg AX, Chow CK, Ackland G, Patel A, Borges FK, Belley-Cote EP, Duceppe E, Spence J, Tandon V, Williams C, Sapsford RJ, Polanczyk CA, Tiboni M, Alonso-Coello P, Faruqui A, Heels-Ansdell D, Lamy A, Whitlock R, LeManach Y, Roshanov PS, McGillion M, Kavsak P, McQueen MJ, Thabane L, Rodseth RN, Buse GAL, Bhandari M, Garutti I, Jacka MJ, Schunemann HJ, Cortes OL, Coriat P, Dvirnik N, Botto F, Pettit S, Jaffe AS and Guyatt GH. Association of Postoperative High-Sensitivity Troponin Levels With Myocardial Injury and 30-Day Mortality Among Patients Undergoing Noncardiac Surgery. JAMA. 2017;317:1642-1651.
- [Background] 1. Halvorsen S, Mehilli J, Cassese S, Hall TS, Abdelhamid M, Barbato E, De Hert S, de Laval I, Geisler T, Hinterbuchner L, Ibanez B, Lenarczyk R, Mansmann UR, McGreavy P, Mueller C, Muneretto C, Niessner A, Potpara TS, Ristic A, Sade LE, Schirmer H, Schupke S, Sillesen H, Skulstad H, Torracca L, Tutarel O, Van Der Meer P, Wojakowski W, Zacharowski K, Group ESCSD, Knuuti J, Kristensen SD, Aboyans V, Ahrens I, Antoniou S, Asteggiano R, Atar D, Baumbach A, Baumgartner H, Bohm M, Borger MA, Bueno H, Celutkiene J, Chieffo A, Cikes M, Darius H, Delgado V, Devereaux PJ, Duncker D, Falk V, Fauchier L, Habib G, Hasdai D, Huber K, Iung B, Jaarsma T, Konradi A, Koskinas KC, Kotecha D, Landmesser U, Lewis BS, Linhart A, Lochen ML, Maeng M, Manzo-Silberman S, Mindham R, Neubeck L, Nielsen JC, Petersen SE, Prescott E, Rakisheva A, Saraste A, Sibbing D, Siller-Matula J, Sitges M, Stankovic I, Storey RF, Ten Berg J, Thielmann M and Touyz RM. 2022 ESC Guidelines on cardiovascular assessment and management of patients undergoing non-cardiac surgery. Eur Heart J. 2022.